CLINICAL TRIAL: NCT06747429
Title: Cardiac Metabolic Reprogramming by a Nutritional Intervention: High Fat Diet for Heart Failure
Brief Title: High Fat Diet for Cardiac Metabolic Reprogramming
Acronym: HF4HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: INSTITUTO DE SALUD CARLOS III (ISCIII) (Unknown); Puerta de Hierro Majadahonda University Hospital (Unknown); Nicole Karam, European Hospital Georges Pompidou, Paris, France (Unknown); Carol Davila University of Medicine and Pharmacy Bucharest (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CARDINNOV; 101095426 (Other Grant/Funding Number: Co-funded by the European Union under the Horizon Europe Framework Programme)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Hearth Failure Secondary to Non-ischemic DCM with Reduced LVEF (≤40%)
Keywords: heart failure; dilated cardiomyopathy; high-fat diet; clinical trial
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated | interventions — Diet, High-Fat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking will be maintained for data analysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High fat diet (Experimental): Patients receiving a high-fat diet
  Interventions: Other: High fat diet
- Control (Active Comparator): Patients receiving a standard diet
  Interventions: Other: Standard diet

INTERVENTIONS:
Other: High fat diet — Weekly isocaloric dietary profile, with total daily energy intake distributed as follows: 70% from fats, primarily sourced from nuts, extra virgin olive oil, avocados, and animal fats from fish and cheese; protein intake of 0.8-1.2 g per kg body weight (10-20%); and the remaining calories from carbohydrates (10-20%).
  Arms: High fat diet
Other: Standard diet — Weekly isocaloric dietary profile, with total daily energy intake distributed as follows: 30% from fats, primarily sourced from nuts, extra virgin olive oil, avocados, and animal fats from fish and cheese; protein intake of 0.8-1.2 g per kg body weight (10-20%); and 50-60% from carbohydrates.
  Arms: Control

SUMMARY:
The heart is a unique organ that performs an incessant work to pump blood throughout the body. For this massive effort, it requires a very high supply of energy. Mitochondria are small components of the cells responsible for the production of energy. To produce energy, mitochondria from cardiac cells can use fuel of different origins (fats, glucose, proteins, etc). In normal circumstances, cardiac mitochondria use preferentially fats since they are more efficient in terms of quantify of energy produced. Recent data from our consortium has demonstrated that if the cardiac mitochondria switch the primary source of fuel (from fats to glucose), this results in a poor performance of the organ, which cannot supply the whole body with enough blood. This is known as heart failure. In experimental models of heart failure, we have demonstrated that a high fat diet is able to reverse the metabolic switch and make the cardiac cells mitochondria use again fats as the primary substrate to produce energy. This translates into a recovery of heart failure. In the present project, we plan to bring this concept to the human setting and perform a pilot clinical study where patients with heart failure are put in a dietary program consisting of high fat diet. The effect of this nutritional approach will be evaluated by state-of-the-art non-invasive imaging technology.

DETAILED DESCRIPTION:
Heart failure (HF) is a progressive condition in which the heart muscle is unable to pump blood effectively to meet the body's needs. It affects millions of people globally and imposes a significant burden on healthcare systems due to its high morbidity, mortality, and economic costs. As the prevalence of HF continues to rise, exploring targeted and innovative treatment strategies is becoming increasingly important.

The heart sustains high energy demands and primarily relies on fatty acids as its energy source in the fasting state, with a smaller contribution from glucose. During the progression of HF, there is a shift in cardiac substrate preference toward increased glucose reliance and reduced fatty acid utilization. Initially considered a protective adaptation against oxygen deficiency and lipotoxicity, this metabolic shift led to suggestions that inhibiting fatty acid oxidation could be a therapeutic strategy for HF. However, more recent evidence indicates that enhancing fatty acid utilization through a high-fat diet may attenuate cardiac dysfunction.

Animal studies have demonstrated that increasing fatty acid utilization can reverse myocardial metabolic alterations and improve cardiac function in models of progressive dilated cardiomyopathy (DCM) with reduced ejection fraction. In one study, the administration of a high-fat diet restored normal myocardial metabolism, resulting in disease regression. Similarly, research using large animal models has shown that high-fat diets can significantly improve left ventricular ejection fraction (LVEF), further supporting the potential benefits of this approach.

In human studies, preliminary findings suggest that lipid-based interventions may acutely improve cardiac function in individuals with HF and reduced LVEF. However, evidence on the long-term efficacy and safety of high-fat dietary patterns in HF management remains limited.

This study aims to compare the effects of a high-fat diet versus a standard diet with a conventional macronutrient composition on non-ischemic DCM with reduced LVEF. The primary objective is to evaluate and compare the impact of a high-fat diet versus a standard diet on LVEF. Secondary objectives include assessing the effects on left ventricular strain, diastolic function, and blood parameters, as well as evaluating the feasibility and degree of adherence to each dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis with HF secondary to non-ischemic DCM with reduced LVEF (≤40%)
* 18 years or older
* informed consent provided

Exclusion Criteria:

* diagnosis of ischemic dilated cardiomyopathy
* recent changes in drug treatment
* significant HF impairment within the past year
* uncontrolled dyslipidemia
* claustrophobia
* presence of a pacemaker or implantable cardiac defibrillator (ICD)
* liver diseases
* life expectancy less than 12 months
* baseline fat intake exceeding 40% of total daily energy intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Changes in left ventricular ejection fraction (LVEF) | At baseline, month 2 and month 4
  Changes in LVEF assessed using cardiac magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Left ventricular strain | At baseline, month 2 and month 4
  Changes in left ventricular strain assessed using cardiac magnetic resonance imaging (MRI)
Diastolic function | At baseline, month 2 and month 4
  Changes in diastolic function assessed using cardiac magnetic resonance imaging (MRI)
White blood cells | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Red blood cells | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Hemoglobin | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Platelets | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Glucose | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
HDL-cholesterol | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
LDL-cholesterol | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Triglycerides | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Electrolytes (sodium, potassium, calcium, magnesium) | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Kidney function (creatinine, urea) | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Vitamins (vitamin B12, 25-OH Vitamin D, folate) | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Albumin | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Iron metabolism (iron, ferritin) | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
Liver function (AST, ALT, γGT) | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures
C-reactive protein | At baseline, month 2 and month 4
  Quantification with standard laboratory procedures

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect participants' privacy.

REFERENCES:
- [Background] Watson WD, Green PG, Lewis AJM, Arvidsson P, De Maria GL, Arheden H, Heiberg E, Clarke WT, Rodgers CT, Valkovic L, Neubauer S, Herring N, Rider OJ. Retained Metabolic Flexibility of the Failing Human Heart. Circulation. 2023 Jul 11;148(2):109-123. doi: 10.1161/CIRCULATIONAHA.122.062166. Epub 2023 May 18. PMID 37199155
- [Background] Stanley WC, Dabkowski ER, Ribeiro RF Jr, O'Connell KA. Dietary fat and heart failure: moving from lipotoxicity to lipoprotection. Circ Res. 2012 Mar 2;110(5):764-76. doi: 10.1161/CIRCRESAHA.111.253104. PMID 22383711
- [Background] Stanley WC, Recchia FA. Lipotoxicity and the development of heart failure: moving from mouse to man. Cell Metab. 2010 Dec 1;12(6):555-6. doi: 10.1016/j.cmet.2010.11.016. PMID 21109186
- [Background] Martinez-Milla J, Galan-Arriola C, Carnero M, Cobiella J, Perez-Camargo D, Bautista-Hernandez V, Rigol M, Solanes N, Villena-Gutierrez R, Lobo M, Mateo J, Vilchez-Tschischke JP, Salinas B, Cusso L, Lopez GJ, Fuster V, Desco M, Sanchez-Gonzalez J, Ibanez B. Translational large animal model of hibernating myocardium: characterization by serial multimodal imaging. Basic Res Cardiol. 2020 Apr 14;115(3):33. doi: 10.1007/s00395-020-0788-0. PMID 32291522
- [Background] Wai T, Garcia-Prieto J, Baker MJ, Merkwirth C, Benit P, Rustin P, Ruperez FJ, Barbas C, Ibanez B, Langer T. Imbalanced OPA1 processing and mitochondrial fragmentation cause heart failure in mice. Science. 2015 Dec 4;350(6265):aad0116. doi: 10.1126/science.aad0116. PMID 26785494
- [Background] Tan Y, Li M, Wu G, Lou J, Feng M, Xu J, Zhou J, Zhang P, Yang H, Dong L, Li J, Zhang X, Gao F. Short-term but not long-term high fat diet feeding protects against pressure overload-induced heart failure through activation of mitophagy. Life Sci. 2021 May 1;272:119242. doi: 10.1016/j.lfs.2021.119242. Epub 2021 Feb 16. PMID 33607155
- [Background] Guo Y, Wang Z, Qin X, Xu J, Hou Z, Yang H, Mao X, Xing W, Li X, Zhang X, Gao F. Enhancing fatty acid utilization ameliorates mitochondrial fragmentation and cardiac dysfunction via rebalancing optic atrophy 1 processing in the failing heart. Cardiovasc Res. 2018 Jun 1;114(7):979-991. doi: 10.1093/cvr/cvy052. PMID 29490017
- [Background] Duda MK, O'Shea KM, Lei B, Barrows BR, Azimzadeh AM, McElfresh TE, Hoit BD, Kop WJ, Stanley WC. Low-carbohydrate/high-fat diet attenuates pressure overload-induced ventricular remodeling and dysfunction. J Card Fail. 2008 May;14(4):327-35. doi: 10.1016/j.cardfail.2007.11.003. PMID 18474346
- [Background] Fillmore N, Mori J, Lopaschuk GD. Mitochondrial fatty acid oxidation alterations in heart failure, ischaemic heart disease and diabetic cardiomyopathy. Br J Pharmacol. 2014 Apr;171(8):2080-90. doi: 10.1111/bph.12475. PMID 24147975
- [Background] Neubauer S. The failing heart--an engine out of fuel. N Engl J Med. 2007 Mar 15;356(11):1140-51. doi: 10.1056/NEJMra063052. No abstract available. PMID 17360992
- [Background] Doenst T, Nguyen TD, Abel ED. Cardiac metabolism in heart failure: implications beyond ATP production. Circ Res. 2013 Aug 30;113(6):709-24. doi: 10.1161/CIRCRESAHA.113.300376. PMID 23989714
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Savarese G, Becher PM, Lund LH, Seferovic P, Rosano GMC, Coats AJS. Global burden of heart failure: a comprehensive and updated review of epidemiology. Cardiovasc Res. 2023 Jan 18;118(17):3272-3287. doi: 10.1093/cvr/cvac013. PMID 35150240